CLINICAL TRIAL: NCT00676455
Title: Computer Assisted Volumetric Analysis of CT-Identified Metastatic Pulmonary Or Hepatic Lesions
Status: Terminated | Type: Observational
Why Stopped: Low participant enrollment, Insufficient findings for data analysis
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-017
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Metastatic Cancer
Keywords: CT Software; MeVis™; Metastatic pulmonary and hepatic lesion growth
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the ability of a new type of CT computer program(MeVis™)to accurately analyze and measure the size and changes in metastatic Liver and Lung tumors. This study will evaluate the data from current CT evaluation methods using the MeVis™ 3-D software.

DETAILED DESCRIPTION:
This is a Pilot Study that will evaluate if metastatic liver and lung tumor measurements made by the MeVis™ software program can provide more accurate information about the size and changes of the tumor compared to the current evaluation method, RECIST(Response Evaluation In Solid Tumors). This study will also collect information about the kind of treatment each subject receives.

Subjects will receive standard of care surveillance CT examinations(a baseline to document tumor size and interval CT exams as indicated by the Oncology Department Protocols); the tumor will be measured according to the current standard-RECIST by Radiology personnel not involved in the study. The CT data will then be analyzed by investigators using the MeVis™ software.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with cancer metastatic to either the liver or lungs
* Subjects Scheduled for regular CT surveillance examinations
* Subjects with life expectancy of at least 6 months

Exclusion Criteria:

* Age <18 years
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects to be recruited from the practice of the Oncology Department. All subjects with hepatic or pulmonary metastatic lesions will be offered the opportunity to participate
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Wald, M.D., Ph.D, Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 100 participants were to be enrolled, with approximately 50 of each type of metastatic disease. 50 participants with metastatic Liver tumors and 50 with metastatic Lung tumors.
Groups:
- Metastatic Lung and Liver Tumor Growth Measurement: This arm of the study will collect information (size and volume changes)of metastatic Lung and Liver tumors
Period: Overall Study
Arm/Group | Metastatic Lung and Liver Tumor Growth Measurement
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metastatic Lung and Liver Tumor Growth Measurement
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: This Study Assessed the Ability of MeVis™ Volumetry Software to Reproducibly Measure the Changes in Metastatic Hepatic and Pulmonary Lesions
Description: Due to the low enrollment for this project the data collected is not sufficient to provide any significant conclusion to the primary outcome hypothesis.
  Due to lack of participants. No significant findings are reported at this time.
Time Frame: As long as treatment is being assessed by CT examinations
Population: Due to low enrollment no analysis was conducted due to the lack of participants.
Arm/Group | Metastatic Lung and Liver Tumor Growth Measurement
Number analyzed (Participants) | 0

2. Secondary Outcome: Tumor Size Will be Measured by CT (by the MeVis Volumetry Software and Correlated With On-going Treatment Plan.
Description: Tumor size will be measured by CT (by the MeVis Volumetry Software and correlated with on-going treatment plan.
  Correlation of the tumor growth with clinical treatment will be assessed. Tumor size will be expressed in volume. Specifically Three dimensional volume Volume of Interest(VOI)will be calculated and correlated with the treatment protocol. Measure = tumor volume.
Time Frame: As long as treatment is being assessed by CT examinations
Population: Due to low enrollment no analysis was conducted due to the lack of participants.
Arm/Group | Metastatic Lung and Liver Tumor Growth Measurement
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Metastatic Lung and Liver Tumor Growth Measurement
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No